CLINICAL TRIAL: NCT05959707
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Monoclonal Antibodies VRC01.23LS, PGT121.414.LS and PGDM1400LS Administered Via Intravenous Infusion in Adults Without HIV
Brief Title: Evaluating the Safety, Tolerability, and Pharmacokinetics of Monoclonal Antibodies in Healthy Participants
Acronym: HVTN143
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Mild Adverse Event related to VRC01.23LS administration was reported.
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 143/HPTN 109; UM1AI068614 (NIH)
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- VRC01.23LS 5 mg/kg (Experimental): VRC01.23LS 5 mg/kg to be administered via intravenous (IV) infusion at Month 0
  Interventions: Biological: VRC01.23LS
- VRC01.23LS 20 mg/kg (Experimental): VRC01.23LS 20 mg/kg to be administered via IV infusion at Month 0
  Interventions: Biological: VRC01.23LS
- VRC01.23LS 40 mg/kg (Experimental): VRC01.23LS 40 mg/kg to be administered via IV infusion at Month 0
  Interventions: Biological: VRC01.23LS
- VRC01.23LS 5 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg (Experimental): VRC01.23LS 5 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg to be administered via IV infusion sequentially in this order at Month 0 and Month 6
  Interventions: Biological: VRC01.23LS; Biological: PGT121.414.LS; Biological: PGDM1400LS
- VRC01.23LS 20 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg (Experimental): VRC01.23LS 20 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg to be administered via IV infusion sequentially in this order at Month 0 and Month 6
  Interventions: Biological: VRC01.23LS; Biological: PGT121.414.LS; Biological: PGDM1400LS
- VRC01.23LS 20 mg/kg + PGT121.414.LS 20 mg/kg+ PGDM1400LS 20 mg/kg (Experimental): VRC01.23LS 20 mg/kg + PGT121.414.LS 20 mg/kg+ PGDM1400LS 20 mg/kg to be administered via IV infusion sequentially in this order at Month 0 and Month 6
  Interventions: Biological: VRC01.23LS; Biological: PGT121.414.LS; Biological: PGDM1400LS
- VRC01.23LS 40 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg (Experimental): VRC01.23LS 40 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg to be administered via IV infusion sequentially in this order at Month 0 and Month 6
  Interventions: Biological: VRC01.23LS; Biological: PGT121.414.LS; Biological: PGDM1400LS
- VRC01.23LS 40 mg/kg + PGT121.414.LS 40 mg/kg + PGDM1400LS 40mg/kg (Experimental): VRC01.23LS 40 mg/kg + PGT121.414.LS 40 mg/kg + PGDM1400LS 40mg/kg to be administered via IV infusion sequentially in this order at Month 0 and Month 6
  Interventions: Biological: VRC01.23LS; Biological: PGT121.414.LS; Biological: PGDM1400LS

INTERVENTIONS:
Biological: VRC01.23LS — VRC01.23LS will be administered IV over approximately 30 to 60 minutes.
Biological: PGT121.414.LS — PGT121.414.LS will be administered IV over approximately 30 to 60 minutes.
  Arms: VRC01.23LS 20 mg/kg + PGT121.414.LS 20 mg/kg+ PGDM1400LS 20 mg/kg; VRC01.23LS 20 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg; VRC01.23LS 40 mg/kg + PGT121.414.LS 40 mg/kg + PGDM1400LS 40mg/kg; VRC01.23LS 40 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg; VRC01.23LS 5 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg
Biological: PGDM1400LS — PGDM1400LS will be administered IV over approximately 30 to 60 minutes.
  Arms: VRC01.23LS 20 mg/kg + PGT121.414.LS 20 mg/kg+ PGDM1400LS 20 mg/kg; VRC01.23LS 20 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg; VRC01.23LS 40 mg/kg + PGT121.414.LS 40 mg/kg + PGDM1400LS 40mg/kg; VRC01.23LS 40 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg; VRC01.23LS 5 mg/kg + PGT121.414.LS 5 mg/kg + PGDM1400LS 5 mg/kg

SUMMARY:
Part A:

The purpose of this part is to study how the body's immune system reacts to a lab-made HIV-1 monoclonal antibody against HIV antigen when given in different doses. The study will also evaluate if the antibody is safe to give to people and does not make them too uncomfortable.

Part B:

The purpose of this part is to study how the body's immune system reacts to a combination of lab-made HIV-1 monoclonal antibodies against HIV antigens when given in different doses. The study also wants to see if the way the antibodies are given affects the immune response.

DETAILED DESCRIPTION:
This study aims to evaluate the safety, tolerability, dose, and PK of VRC01.23LS administered IV and in combination with PGDM1400LS, a V2-apex-targeting mAb, and PGT121.414.LS, a V3-glycan-targeting mAb.

There are 2 parts to this study: Part A and Part B.

In Part A, 15 participants will be randomly assigned to test one study antibody at different doses.

After we see the results from Part A, we will decide whether or not to do Part B of the study.

In Part B, 62 participants will be randomly assigned to test a combination of 3 study antibodies, including the one tested in Part A.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 through 50 years
2. Access to a participating CRS and willingness to be followed for the planned duration of the study
3. Ability and willingness to provide informed consent
4. Assessment of understanding (AoU): volunteer demonstrates understanding of this study and completes a questionnaire prior to first study-product administration with verbal demonstration of understanding of all questionnaire items answered incorrectly
5. Agrees not to enroll in another study of an investigational research agent until completion of the last required protocol clinic visit.
6. Good general health as shown by medical history, physical exam, and screening laboratory tests
7. Willingness to receive HIV test results
8. Willingness to discuss HIV acquisition and amenable to HIV risk-reduction counseling.
9. Assessed by the clinic staff as having a low likelihood of HIV acquisition and is committed to avoid behaviors associated with a higher likelihood of acquiring HIV through the last required protocol clinic visit.
10. Hemoglobin

    * ≥ 11.0 g/dL for AFAB volunteers
    * ≥ 13.0 g/dL for AMAB volunteers and transgender men who have been on hormone therapy for more than 6 consecutive months
    * ≥ 12.0 g/dL for transgender women who have been on hormone therapy for more than 6 consecutive months
    * For transgender volunteers who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on their sex assigned at birth
11. White blood cell (WBC) count = 2,500 to 12,000 cells/mm3
12. WBC differential either within institutional normal range or with site clinician approval
13. Platelets = 125,000 to 550,000 cells/mm3
14. Chemistry panel: alanine aminotransferase (ALT) < 1.25 times the institutional upper limit of normal (ULN) (ie, < 1.25 times the reference range upper limit) and creatinine < 1.1 times the institutional ULN (ie, < 1.1 times the reference range upper limit)
15. Negative HIV-1 and -2 blood test: Sites may use locally available assays that have been approved by HVTN and HPTN Laboratory Operations
16. Negative Hepatitis B surface antigen (HBsAg)
17. Negative anti-Hepatitis C virus Abs (anti-HCV) or negative HCV PCR if the anti-HCV is positive
18. Negative or trace urine protein
19. AFAB volunteers or volunteers who were intersex at birth and are capable of becoming pregnant (hereafter referred to as "persons of pregnancy potential"): negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test(s) performed within 48 hours prior to initial study-product administration. Persons who are NOT of pregnancy potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records) are not required to undergo pregnancy testing.
20. Persons of pregnancy potential must:

    * Agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol visit. Effective contraception is defined as using one of the following methods:

      * Condoms (internal and external) with or without a spermicide,
      * Diaphragm or cervical cap with spermicide,
      * Intrauterine device (IUD),
      * Hormonal contraception,
      * Tubal ligation, or
      * Any other contraceptive method approved by the HVTN 143/HPTN 109 PSRT
      * Successful vasectomy in any AMAB partner (considered successful if a volunteer reports that an AMAB partner has [1] documentation of azoospermia by microscopy or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy); or,
    * Not be of pregnancy potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy or bilateral oophorectomy; or,
    * Be sexually abstinent.
21. AFAB volunteers or who were intersex at birth must also agree not to seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks until after the last required protocol clinic visit

Exclusion Criteria:

1. Weight < 35 kg or > 115 kg
2. Blood products received within 120 days before first study-product administration, unless eligibility for earlier enrollment is determined by the HVTN 143/HPTN 109 PSRT
3. Investigational research agents received within 30 days before first study-product administration
4. Intent to participate in another study of an investigational research agent or any other study that requires non-Network HIV Ab testing during the planned duration of the HVTN 143/HPTN 109 study
5. Pregnant or breastfeeding
6. HIV vaccine(s) received in a prior HIV vaccine trial. Volunteers who have received control/placebo in an HIV vaccine trial are not excluded from HVTN 143/HPTN 109.
7. SARS-CoV-2 vaccine(s) received within 7 days prior to HVTN 143/HPTN 109 enrollment or planned within 7 days after enrollment.
8. Jynneos vaccine for MPOX received within 14 days prior to enrollment or planned within 14 days after enrollment.
9. ACAM2000 vaccine for MPOX received within 28 days prior to enrollment or, if ACAM2000 was received more than 28 days prior to enrollment, vaccination scab still present; or planned within 14 days after enrollment
10. Receipt of humanized or human mAbs, whether licensed or investigational.
11. Previous receipt of mAbs targeting HIV (eg, cap256, VRC01, VRC01LS, VRC07-523LS, PGDM1400, PGDM1400LS, PGT121, PGT121.414.LS)
12. Immunosuppressive medications received within 30 days before first study-product administration (not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatological condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses < 20 mg/day and length of therapy < 14 days, but completed at least 7 days prior to first infusion)
13. Serious adverse reactions to VRC01.23LS, PGDM1400LS, or PGT121.414.LS formulation components, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
14. Immunoglobulin received within 60 days before first study-product administration (for mAb, see criterion 10 above)
15. Autoimmune disease (not exclusionary: volunteer with mild, stable, and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the CRS investigator, is likely not subject to exacerbation and likely not to complicate solicited and unsolicited AE assessments)
16. Immunodeficiency
17. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * Symptoms consistent with COVID-19 or known SARS-CoV-2 acquisition,
    * A process that would affect the immune response,
    * A process that would require medication that affects the immune response,
    * Any contraindication to repeated infusions or blood draws, including inability to establish venous access,
    * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
    * A condition or process (eg, chronic urticaria or recent injection or infusion with evidence of residual inflammation) for which signs or symptoms could be confused with reactions to the study product, or
    * Any condition specifically listed among the exclusion criteria.
18. Any medical, psychiatric, or skin condition (eg, tattoos) or occupational responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety or solicited AEs, or a participant's ability to give informed consent.
19. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses, ongoing risk for suicide, or history of suicide attempt within the past 3 years.
20. Current anti-tuberculosis (TB) therapy
21. Asthma other than mild, well-controlled asthma (symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program [NAEPP] Expert Panel report).

    Exclude a volunteer who:
    * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily; or
    * Uses moderate/high-dose, inhaled corticosteroids; or
    * In the past year, has had either of the following:

      * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
      * Emergency care, urgent care, hospitalization, or intubation for asthma.
22. Diabetes mellitus type 1 or type 2 (not exclusionary: type-2 cases controlled with diet alone or a history of isolated gestational diabetes)
23. Hypertension

    * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
    * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
24. Bleeding disorder diagnosed by a clinician (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
25. Malignancy (not exclusoinary: volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
26. Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
27. Asplenia: any condition resulting in the absence of a functional spleen
28. History of generalized urticaria, angioedema, or anaphylaxis (not exclusionary: angioedema or anaphylaxis to a known trigger with at least 5 years since last reaction to demonstrate satisfactory avoidance of trigger)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Estimated)
Dates: Start 2024-08-14 (Estimated); Primary Completion 2025-01-14 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Number of Local and systemic solicited AEs | Through 6 months
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Number of unsolicited AEs, and SAEs | Through 6 months
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Serum concentrations of PGT121.414.LS | Through 6 months
  Measured using quantitative immunoassay
Serum concentrations of VRC01.23LS | Through 6 months
  Measured using quantitative immunoassay
Serum concentrations of PGDM1400LS | Through 6 months
  Measured using quantitative immunoassay
Magnitude of serum neutralizing activity measured with mAb-specific Env-pseudotyped viruses in TZM-bl cells | Through 6 months
  Measured using HIV-1-specific nAb assays

SECONDARY OUTCOMES:
Serum concentrations of VRC01.23LS | Through 8 months
  Measured using quantitative immunoassay
Serum concentrations of PGT121.414.LS | Through 8 months
  Measured using quantitative immunoassay
Serum concentrations of PGDM1400LS | Through 8 months
  Measured using quantitative immunoassay
Magnitude of serum neutralizing activity measured with Env-pseudotyped viruses in TZM-bl cells | Through 8 months
  Measured using HIV-1-specific nAb assays
Magnitude of neutralizing activity against a panel of Env-pseudotyped reference viruses in TZM-bl cells | Through 8 months
  Measured using HIV-1-specific nAb assays
Serum concentrations of ADA titer | Through 8 months
  Measured using quantitative immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Scott, Study Chair — Bridge HIV; Cynthia Gay, Study Chair — University of North Carolina
Locations (8):
- South Africa (8):
  - Groote Schuur HIV CRS, Cape Town, Western Cape
  - Emavundleni CRS, Klipfontein, Western Cape
  - CAPRISA eThekwini CRS, Durban
  - Soweto HPTN CRS, Johannesburg
  - Ward 21 CRS, Johannesburg
  - Klerksdorp CRS, Klerksdorp
  - Isipingo CRS, KwaZulu
  - Soshanguve, Soshanguve